CLINICAL TRIAL: NCT04738500
Title: Postoperative Analgesic Efficacy of Pericapsular Nerve Group Block (PENG) Block for Knee Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bora Bilal (Other)
Responsible Party: Sponsor-Investigator, Bora Bilal, Principal investigator, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG Block (Active Comparator): PENG Block combinate with PCA
  Interventions: Procedure: PENG Block combinated with PCA
- CONTROL (Sham Comparator): PCA
  Interventions: Procedure: PCA

INTERVENTIONS:
Procedure: PENG Block combinated with PCA — After spinal anesthesia PENG block will be performed
  Other Names: PCA
  Arms: PENG Block
Procedure: PCA — PCA will be applied after surgery
  Arms: CONTROL

SUMMARY:
Pericapsular nerve group block (PENG) has been deemed as a safe and effective regional technique for postoperative pain after knee arthroscopy.

DETAILED DESCRIPTION:
Pericapsular nerve group block(PENG) has been deemed as a safe and effective regional technique for postoperative pain after knee artroscopy. Blockade of the branches of the femoral and obturator nerves that provide innervation to any structures distal enough to be useful in knee.

ELIGIBILITY:
Inclusion Criteria:

* Patients agreed to receive PENG block
* Knee arthroscopy

Exclusion Criteria:

* Other kinds of knee surgery
* Patients refuse to receive PENG block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
First analgesic demand | 24 Hours
  The time interval from PENG blocks to the first analgesic demand.

SECONDARY OUTCOMES:
Opioid consumption | 24 Hours
  Total opioid analgesic consumption
Numeric Rating Scale | 24 Hours
  The maximum score on a 10cm numeric rating scale: (0 to 10cm) (0 = no pain, 10 = worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- KSU Faculty of Medicine Research Hospital, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No